CLINICAL TRIAL: NCT06550063
Title: HER2 Status in Esophagogastric Adenocarcinoma and Its Associations With Patient's Clinicopathological Outcomes
Acronym: HERA
Status: Recruiting | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Nicola Raftery, Principal investigator, Dr, St. James's Hospital, Ireland
Other Study IDs: HERA001
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Esophagus Cancer; Gastric Cancer; HER2-positive Cancer; HER2-low Cancer
Keywords: Esophageal cancer; Gastric cancer; HER2-positive cancer; HER2-low cancer; Targeted treatment
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Targeted therapies offer promise to improve oncologic outcomes in esophagogastric adenocarcinoma (EGA). The landmark 'Trastuzumab for gastric cancer (ToGA)' trial established the therapeutic value of Human Epidermal Growth Factor Receptor 2 (HER2) directed therapy in advanced gastric and esophagogastric junction adenocarcinoma, setting a standard of care. Further studies, such as DESTINY-gastric01 and DESTINY-gastric02, have demonstrated the efficacy of antibody-drug conjugates (ADCs) targeting HER2-positive gastric and junctional tumours. The use of HER2-directed therapies in the curative intent setting has more recently been evaluated with favourable outcomes in phase II studies. However, data regarding the prevalence and prognostic significance of HER2 overexpression among patients undergoing treatment with curative intent are limited. Furthermore, few studies have evaluated the clinical significance of intratumoural and tumour-metastatic heterogeneity of HER2 expression, and the finding of HER2-low, in this context, which may have important implications for implementation of neoadjuvant targeted therapies in future. While limited single centre series have evaluated the clinicopathologic significance of HER2 status in EGA, no previous international multicentre study of this nature has been reported.

The goal of this international, multi-center, retrospective observational study is to elucidate the prevalence and clinical significance of HER2 expression in patients with EGA across different regions globally. The study also aims to assess the clinical significance of HER2 heterogeneity in a large, international cohort of patients with EGA, and its association with clinicopathological outcomes in patients with advanced and recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed EGA from 2000 to April 2024 across all stages of disease
* Primary tumour HER2 status tested as routine in all patients with EGA
* Patients aged 18 years or over

Exclusion Criteria:

- Patients with esophageal squamous cell carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a multi-center, retrospective, international cohort study including a population of patients diagnosed with EGA from 2000 to April 2024 across all stages of disease with primary tumour routinely tested for HER2 status.
Sampling Method: Probability Sample
Enrollment: 2188 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Geographical variation in HER2 status | 2000 - 2024

SECONDARY OUTCOMES:
Clinical TNM stage | 2000 - 2024
Overall survival | 2000 - 2024

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MBBCh,MD, Principal Investigator — Trinity St James Cancer Institute
Locations (1):
- Trinity St James Cancer Institute, Dublin, Leinster, Ireland